CLINICAL TRIAL: NCT06702397
Title: Preliminary Results of Microsurgical Testicular Exploration for Sperm Retrieval in Azoospermic Patients: A Randomized Controlled Trial Comparing Operating Microscope vs. Surgical Loupes
Brief Title: TeSE (Testicular Sperm Extraction) in Azoospermic Patients: m-TeSE vs. l-TeSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Federica Peretti (Unknown); Ilaria Ferro (Unknown); Natalia Plamadeala (Unknown); Martina Scavone (Unknown); Luca Boeri (Unknown); Marco Falcone (Unknown); Lorenzo Cirigliano (Unknown); Valentina Parolin (Unknown); Emanuele Zupo (Unknown); Paolo Gontero (Unknown)
Responsible Party: Principal Investigator, Mirko Preto, Doctor Mirko Preto, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202/2022
Record Dates: First submitted 2024-11-03; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Azoospermia, Nonobstructive
MeSH Terms: conditions — Azoospermia, Nonobstructive

STUDY DESIGN:
Intervention Model Description: Randomized multi-center controlled trial comparing microsurgical-assisted testicular sperm extraction (m-TeSE - Group A) and testicular sperm extraction performed with surgical loupes (l-TeSE - Group B) in adult males with non-obstructive azoospermia (NOA) in terms of surgical outcomes and sperm retrieval rates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microsurgical-assisted testicular sperm extraction (m-TeSE) - Group A (Active Comparator): A longitudinal incision of 3cm was made along the scrotal raphe using a scalpel. Surgical dissection proceeded layer by layer. The testis was separated from the surrounding dartos and luxated outside the scrotal sac. A longitudinal incision was made in the tunica vaginalis to allow complete exposure of the tunica albuginea. Two Vicryl 2-0 traction sutures were placed 0.5 cm cranially and caudally to the testicular equatorial line, which was subsequently incised with a scalpel for 3/4 of the testicular circumference. In M-TESE, through the operating microscope, a direct examination of the testicular parenchyma was performed under magnification (20-25x). Multiple testicular specimens were excised. The same procedure is performed on the contralateral side, where instead of the operating microscope, the surgeon uses surgical loupes for magnification (3.5 - 5x).
  Interventions: Device: Microscope
- Testicular sperm extraction performed with surgical loupes (l-TeSE) - Group B (Active Comparator): A longitudinal incision of 3cm was made along the scrotal raphe using a scalpel. Surgical dissection proceeded layer by layer. The testis was separated from the surrounding dartos and luxated outside the scrotal sac. A longitudinal incision was made in the tunica vaginalis to allow complete exposure of the tunica albuginea. Two Vicryl 2-0 traction sutures were placed 0.5 cm cranially and caudally to the testicular equatorial line, which was subsequently incised with a scalpel for 3/4 of the testicular circumference. In M-TESE, through the operating microscope, a direct examination of the testicular parenchyma was performed under magnification (20-25x). Multiple testicular specimens were excised. The same procedure is performed on the contralateral side, where instead of the operating microscope, the surgeon uses surgical loupes for magnification (3.5 - 5x).
  Interventions: Device: Surgical loupes

INTERVENTIONS:
Device: Microscope — The microscope provides a direct examination of the testicular parenchyma at 20-25x magnification.
  Arms: Microsurgical-assisted testicular sperm extraction (m-TeSE) - Group A
Device: Surgical loupes — Surgical loupes offer magnification of 3.5-5x.
  Arms: Testicular sperm extraction performed with surgical loupes (l-TeSE) - Group B

SUMMARY:
The aim of the study is to compare surgical outcomes (intra and post-operative complications) and sperm retrieval rates between conventional microsurgical-assisted testicular sperm extraction (m-TeSE - Group A) and testicular sperm extraction performed with surgical loupes (l-TeSE - Group B) in adult males with non-obstructive azoospermia.

DETAILED DESCRIPTION:
Objective: To compare surgical outcomes and sperm retrieval rates (SRR) between conventional microsurgical-assisted testicular sperm extraction (m-TeSE - Group A) and testicular sperm extraction performed with surgical loupes (l-TeSE - Group B) in adult males with non-obstructive azoospermia (NOA). A multicentric prospective randomized trial was conducted from March 2022. Adult males with NOA without genetic alterations who agreed to participate in the study and signed the required informed consent were enrolled. SRR, intra and post-operative complications (according to Clavien-Dindo classification), hormonal profile tchanges were considered as outcomes during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult males
* Diagnosis of non obstructive azoospermia who required m-TeSE.

Exclusion Criteria:

* Absence of signed written informed consent
* Age < 18 years
* Obstructive azoospermia
* Genetic anomalies (e.g., Klinefelter syndrome, Kallmann syndrome, Y chromosome microdeletions, CFTR mutations)
* Previous testicular biopsies/surgical sperm retrieval
* Personal history of malignant testicular tumor
* Unilateral cryptorchidism
* Varicocele
* Previous chemotherapy/radiotherapy treatments
* Monorchidism

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Positive sperm retrieval | immediately after the surgery
  Number of sperm retrieval
Histology | immediately after the surgery
  Normal testicular biopsy or Hypospermatogenesis or Germ cell arrest or Sertoli cell-only syndrome or Seminiferous tubule hyalinization or CIS or Immature testis
Johnsen score | immediately after the surgery
  Number according to Johnsen score
Sperm vials stored | immediately after the surgery
  Number

SECONDARY OUTCOMES:
Operative time | immediately after the surgery
  Minutes
Complications | through study completion, an average of 1 year
  Clavien dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Molinette - AOU Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen ML, Buncke GM, Turek PJ. Narrative review of the history of microsurgery in urological practice. Transl Androl Urol. 2021 Apr;10(4):1780-1791. doi: 10.21037/tau-20-1441. PMID 33968665
- [Background] Bernie AM, Mata DA, Ramasamy R, Schlegel PN. Comparison of microdissection testicular sperm extraction, conventional testicular sperm extraction, and testicular sperm aspiration for nonobstructive azoospermia: a systematic review and meta-analysis. Fertil Steril. 2015 Nov;104(5):1099-103.e1-3. doi: 10.1016/j.fertnstert.2015.07.1136. Epub 2015 Aug 8. PMID 26263080
- [Background] Flannigan R, Bach PV, Schlegel PN. Microdissection testicular sperm extraction. Transl Androl Urol. 2017 Aug;6(4):745-752. doi: 10.21037/tau.2017.07.07. PMID 28904907
- [Background] Li H, Chen LP, Yang J, Li MC, Chen RB, Lan RZ, Wang SG, Liu JH, Wang T. Predictive value of FSH, testicular volume, and histopathological findings for the sperm retrieval rate of microdissection TESE in nonobstructive azoospermia: a meta-analysis. Asian J Androl. 2018 Jan-Feb;20(1):30-36. doi: 10.4103/aja.aja_5_17. PMID 28361811
- [Background] Pozzi E, Raffo M, Negri F, Boeri L, Sacca A, Belladelli F, Cilio S, Ventimiglia E, d'Arma A, Pagliardini L, Vigano P, Pontillo M, Luciano R, Colecchia M, Montorsi F, Alfano M, Salonia A. Anti-Mullerian hormone predicts positive sperm retrieval in men with idiopathic non-obstructive azoospermia-findings from a multi-centric cross-sectional study. Hum Reprod. 2023 Aug 1;38(8):1464-1472. doi: 10.1093/humrep/dead125. PMID 37322566
- [Background] Tournaye H, Liu J, Nagy PZ, Camus M, Goossens A, Silber S, Van Steirteghem AC, Devroey P. Correlation between testicular histology and outcome after intracytoplasmic sperm injection using testicular spermatozoa. Hum Reprod. 1996 Jan;11(1):127-32. doi: 10.1093/oxfordjournals.humrep.a019004. PMID 8671174
- [Background] Boeri L, Palmisano F, Preto M, Sibona M, Capogrosso P, Franceschelli A, Ruiz-Castane E, Sarquella-Geli J, Bassas-Arnau L, Scroppo FI, Sacca A, Gentile G, Falcone M, Timpano M, Ceruti C, Gadda F, Trost L, Colombo F, Rolle L, Gontero P, Montorsi F, Sanchez-Curbelo J, Salonia A, Montanari E. Sperm retrieval rates in non-mosaic Klinefelter patients undergoing testicular sperm extraction: What expectations do we have in the real-life setting? Andrology. 2020 May;8(3):680-687. doi: 10.1111/andr.12767. Epub 2020 Feb 16. PMID 31999885
- [Background] Ostad M, Liotta D, Ye Z, Schlegel PN. Testicular sperm extraction for nonobstructive azoospermia: results of a multibiopsy approach with optimized tissue dispersion. Urology. 1998 Oct;52(4):692-6. doi: 10.1016/s0090-4295(98)00322-7. PMID 9763095
- [Background] Pozzi E, Boeri L, Capogrosso P, Palmisano F, Preto M, Sibona M, Franceschelli A, Ruiz-Castane E, Sarquella-Geli J, Bassas-Arnau L, Scroppo FI, Gentile G, Falcone M, Timpano M, Ceruti C, Gadda F, Colombo F, Rolle L, Gontero P, Montorsi F, Sanchez-Curbelo J, Montanari E, Salonia A. Rates of hypogonadism forms in Klinefelter patients undergoing testicular sperm extraction: A multicenter cross-sectional study. Andrology. 2020 Nov;8(6):1705-1711. doi: 10.1111/andr.12843. Epub 2020 Jul 3. PMID 32558292
- [Background] Vieira M, Bispo de Andrade MA, Santana-Santos E. Is testicular microdissection the only way to retrieve sperm for non-obstructive azoospermic men? Front Reprod Health. 2022 Aug 23;4:980824. doi: 10.3389/frph.2022.980824. eCollection 2022. PMID 36303631
- [Background] Serletti JM, Deuber MA, Guidera PM, Reading G, Herrera HR, Reale VF, Wray RC Jr, Bakamjian VY. Comparison of the operating microscope and loupes for free microvascular tissue transfer. Plast Reconstr Surg. 1995 Feb;95(2):270-6. doi: 10.1097/00006534-199502000-00006. PMID 7824606
- [Background] Boeri L, Bebi C, Dente D, Greco E, Turetti M, Capece M, Cocci A, Cito G, Preto M, Pescatori E, Ciampaglia W, Scroppo FI, Falcone M, Ceruti C, Gadda F, Franco G, Deho F, Palmieri A, Rolle L, Gontero P, Montorsi F, Montanari E, Salonia A. Outcomes and predictive factors of successful salvage microdissection testicular sperm extraction (mTESE) after failed classic TESE: results from a multicenter cross-sectional study. Int J Impot Res. 2022 Dec;34(8):795-799. doi: 10.1038/s41443-021-00487-8. Epub 2021 Nov 6. PMID 34743195
- [Background] Falcone M, Boeri L, Timpano M, Cirigliano L, Preto M, Russo GI, Peretti F, Ferro I, Plamadeala N, Gontero P. Combined Trifocal and Microsurgical Testicular Sperm Extraction Enhances Sperm Retrieval Rate in Low-Chance Retrieval Non-Obstructive Azoospermia. J Clin Med. 2022 Jul 13;11(14):4058. doi: 10.3390/jcm11144058. PMID 35887821
- [Background] Schlegel PN, Su LM. Physiological consequences of testicular sperm extraction. Hum Reprod. 1997 Aug;12(8):1688-92. doi: 10.1093/humrep/12.8.1688. PMID 9308794
- [Background] Schoysman R, Vanderzwalmen P, Nijs M, Segal L, Segal-Bertin G, Geerts L, van Roosendaal E, Schoysman D. Pregnancy after fertilisation with human testicular spermatozoa. Lancet. 1993 Nov 13;342(8881):1237. doi: 10.1016/0140-6736(93)92217-h. No abstract available. PMID 7901551
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Zhao H, Xu J, Zhang H, Sun J, Sun Y, Wang Z, Liu J, Ding Q, Lu S, Shi R, You L, Qin Y, Zhao X, Lin X, Li X, Feng J, Wang L, Trent JM, Xu C, Gao Y, Zhang B, Gao X, Hu J, Chen H, Li G, Zhao J, Zou S, Jiang H, Hao C, Zhao Y, Ma J, Zheng SL, Chen ZJ. A genome-wide association study reveals that variants within the HLA region are associated with risk for nonobstructive azoospermia. Am J Hum Genet. 2012 May 4;90(5):900-6. doi: 10.1016/j.ajhg.2012.04.001. Epub 2012 Apr 26. PMID 22541561
- [Background] Jarow JP, Espeland MA, Lipshultz LI. Evaluation of the azoospermic patient. J Urol. 1989 Jul;142(1):62-5. doi: 10.1016/s0022-5347(17)38662-7. PMID 2499695